CLINICAL TRIAL: NCT03282916
Title: Anti-viral Therapy in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Devangere P. Devanand, Professor of Clinical Psychiatry and Neurology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAV1800; R01AG055422 (NIH); NYSPI 7537 (Other: New York State Psychiatric Institute)
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Results first posted 2025-09-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease; Herpes Simplex 1; Herpes Simplex 2
Keywords: Valacyclovir; Anti-viral treatment
MeSH Terms: conditions — Alzheimer Disease | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Valacyclovir (Active Comparator): The oral valacyclovir will be distributed in 500mg caplets. Patients will take 8 caplets per day.
  Interventions: Drug: Valacyclovir
- Placebo (Placebo Comparator): The oral placebo (sugar pill) will be distributed in 500mg caplets. Patients will take 8 caplets per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valacyclovir — Valacyclovir hydrochloride 500mg caplet
  Other Names: Valtrex
  Arms: Valacyclovir
Drug: Placebo — Placebo sugar pill 500mg caplet
  Arms: Placebo

SUMMARY:
Anti-viral therapy in Alzheimer's disease will investigate the efficacy of treating patients with mild Alzheimer's disease with the U.S.A marketed generic anti-viral drug Valtrex (valacyclovir, 500mg oral tablet). Valacyclovir, titrated to 4 grams per day, repurposed to treat Alzheimer's disease, will be compared to matching placebo in the treatment of 130 mild AD patients (65 valacyclovir, 65 placebo) who test positive for herpes simplex virus-1 (HSV1) or herpes simplex virus-2 (HSV2). The study will be a randomized, double-blind, 18-month Phase II proof of concept trial.

DETAILED DESCRIPTION:
Many viruses are latent for decades before being reactivated in the brain by stress, immune compromise, or other factors. After the initial oral infection, herpes simplex virus-1 (HSV1) becomes latent in the trigeminal ganglion and can later enter the brain via retrograde axonal transport, often targeting the temporal lobes.

HSV1 can also enter the brain via olfactory neurons directly. HSV1 (oral herpes) and HSV2 (genital herpes) are known to trigger amyloid aggregation and their DNA is commonly found in amyloid plaques. Anti-HSV drugs reduce Aβ and p-tau accumulation in brains of infected mice. HSV1 reactivation is associated with tau hyperphosphorylation in mice and may play a role in tau propagation across neurons. In humans, recurrent reactivation with newly produced HSV1 particles, 'drop by drop,' may produce neuronal damage and eventually lead to neurodegeneration and Alzheimer's disease (AD) pathology, partly due to effects on amyloid and tau. Clinical studies show cognitive impairment in HSV seropositive patients in different patient groups and in healthy adults, and antiviral treatments show robust efficacy against peripheral HSV infection. The study team will conduct the first-ever clinical trial to directly address the long-standing viral etiology hypothesis of AD which posits that viruses, particularly the very common HSV1 and HSV2, may be etiologic or contribute to the pathology of AD. In patients with mild AD who test positive for serum antibodies to HSV1 or HSV2, the generic antiviral drug valacyclovir, repurposed as an anti-AD drug, will be compared at oral doses of 4 grams per day, to matching placebo in the treatment of 130 patients (65 valacyclovir, 65 placebo) in a randomized, double-blind, 78-week Phase II proof of concept trial. Patients treated with valacyclovir are hypothesized to show smaller decline in cognition and functioning compared to placebo, and, using 18F-Florbetapir PET imaging, to show less amyloid accumulation than placebo over the 78-week trial. Through the use of tau PET imaging with the tracer 18F-MK-6240 at baseline and 78 weeks, patients treated with valacyclovir are hypothesized to show smaller increases in 18F-MK-6240 binding than patients treated with placebo from baseline to 78 weeks. Apolipoprotein E genotype at baseline, as well as changes in cortical thinning on structural MRI, olfactory identification deficits, and antiviral antibody titers from baseline to 78 weeks, will be evaluated in exploratory analyses. In patients who agree to lumbar puncture, plasma and CSF acyclovir will be assayed to establish the degree of CNS penetration of valacyclovir in mild AD, and the investigators will obtain CSF Aβ42, tau, p-tau for subset exploratory analyses with changes in outcome measures. If this trial is successful, the investigators will apply for funding to conduct a larger, multicenter, Phase III study using a study design that will be informed by the results of this Phase II trial. This innovative Phase II proof of concept trial clearly has exceptionally high reward potential for the treatment of AD.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females. Females must be postmenopausal defined as 12 consecutive months without menstruation. Patient Report
2. Diagnosis of probable AD by NIA clinical diagnostic criteria. Physician Evaluation
3. Folstein Mini Mental State (MMSE) score 18 to 28 (inclusive) out of 30. Neuropsychological Evaluation
4. Clinical Dementia Rating (CDR) score of 1 (mild dementia). Physician Evaluation
5. A family member or other individual who is in contact with the patient and consents to serve as informant during the study Patient Report
6. Patient retains capacity to consent for him/herself or retains the capacity to identify a surrogate who will consent on his/her behalf. Patient Report
7. At screening, patients must test positive for serum antibodies to HSV1 or HSV2. Patients that test equivocal (index between 0.90-1.09; < 0.90 is negative and > 1.09 is positive) will repeat the test within 6 weeks at a repeat visit. If the results are negative at the second test, the patient will not enter the study. If the results are equivocal or positive at the second test (first test was equivocal), we will enroll the patient in the study because "equivocal" indicates the presence of antibodies that do not reach the minimum threshold.
8. Use of cholinesterase inhibitors and memantine, and concomitant psychotropic medications (other than high dose benzodiazepines), will be permitted throughout the trial. Doses of these medications will need to be stable for at least 1 month prior to study entry. Any changes to the medication will be documented in the participant research chart. Medications given for other medical reasons, e.g., anti-diabetic or antihypertensive medications, will not be altered for the purposes of this trial and the patient's primary physician may adjust such medications as medically indicated throughout the trial. Details of concomitant medication use will be documented at all visits and will be available for statistical analysis.
9. For patients diagnosed with Mild Cognitive Impairment and CDR score of 0.5 ( questionable dementia), if these patients have biomarkers of AD neuropathology with either a positive amyloid PET scan, positive fluorodeoxyglucose (FDG) PET scan of the brain, or positive findings for AD in CSF ( low ABeta42 and high tau, p-tau protein levels) they will be eligible for the study. This applies to patients who already had an amyloid PET scan, FDG PET scan of the brain, or lumbar puncture, prior to recruitment into the protocol.

Physical Evaluation

Exclusion Criteria:

1. Caregiver is unwilling or unable, in the opinion of the investigator, to comply with study instructions. Physician Evaluation
2. Patient has dementia predominantly of non-Alzheimer's type, including vascular dementia, frontotemporal dementia, Lewy body dementia, substance-induced dementia. Physician Evaluation
3. Modified Hachinski scale score greater than 4. Physician Evaluation
4. Current clinical diagnosis of schizophrenia, schizoaffective disorder, other psychosis, bipolar disorder or current major depression by DSM-5 criteria. Prior history of major depression will not be exclusionary (25% of older adults have a lifetime history of major depression). Physician Evaluation
5. Active suicidal intent or plan based on clinical assessment. Physician Evaluation
6. Current or recent (past 6 months) alcohol or substance use disorder (DSM-5 criteria). Physician Evaluation
7. Current diagnosis of other major neurological disorders, including Parkinson's disease, multiple sclerosis, CNS infection, Huntington's disease, and amyotrophic lateral sclerosis. Physician Evaluation
8. Clinical stroke with residual neurological deficits. MRI findings of cerebrovascular disease (small infarcts, lacunes, periventricular disease) in the absence of clinical stroke with residual neurological deficits will not lead to exclusion. Physician Evaluation
9. Acute, severe, unstable medical illness. For cancer, patients with active illness or metastases in the last 12 months will be excluded, but past history of successfully treated cancer will not lead to exclusion. Physician Evaluation
10. Sitting blood pressure > 160/100 mm Hg. Physician Evaluation
11. Renal failure as determined by an estimated Glomerular Filtration Rate (GFR) < 44 ml/min/1.73m2 (see 4.3.b.). Physician Evaluation/ Laboratory Report
12. Serum vitamin B12 levels below the normal range. Physician Evaluation/ Laboratory Report
13. Patients with thrombotic thrombocytopenic purpura/hemolytic uremic syndrome will be excluded. Physician Evaluation
14. Use of benzodiazepines in lorazepam equivalent doses equal to or greater than 2 mg daily. Physician Evaluation
15. For patients consenting to lumbar puncture (40% of sample), this procedure will be conducted if there is no lower spinal malformation or other contraindication to lumbar puncture. Physician Evaluation
16. For MRI, metal implants and pacemaker, and claustrophobia such that the patient refuses MRI. In the investigators' experience, these exclusions occur in less than 5% of patients with mild AD. MRI is required for VALAD. Patient Report/ Physician Evaluation
17. Radiation exposure in the prior 12 months that, together with 18F-Florbetapir and 18F--MK-6240 PET, will be above the FDA annual radiation exposure threshold. This will be determined through study staff ( i.e. Principal Investigator, Study Physician) discussion with potential subjects at Screening, documenting inquiry about radiation history. If there is any history of additional radiation exposure in the past year; it will be reviewed with PET Center staff for their approval before proceeding. The combined radiation exposure from the maximum doses used for 18F-Florbetapir and 18F-MK- 6240 is within the FDA limits for annual radiation exposure and the second scan in each patient will be done 18 months after the initial PET scan (for both radioligands). Patient Report/Physician Evaluation
18. Severe vision or hearing impairment that would prevent the participant from performing the psychometric tests accurately. This will be a clinical determination by the study physician without formal testing or audiometry Physician Evaluation
19. Olfaction component: current upper respiratory infection (patient tested as soon as this improves), current smoker > 1 pack daily (past smoking has been shown not to affect UPSIT scores, UPSIT score < 12/40 (10 out of 40 is scored by chance in this multiple-choice test) indicating congenital anosmia. In the investigators' experience, less than 3% of cases are excluded for having one or more of these exclusionary criteria. If a patient is excluded from the olfaction component, the patient will still be eligible for the main protocol and all other study procedures. Patient Report/Physician Evaluation

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davangere Devanand, MD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Banner Alzheimer's Institute (BAI), Phoenix, Arizona
  - New York University School of Medicine, New York, New York
  - New York State Psychiatric Institute, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Devanand DP, Wisniewski T, Razlighi Q, Qian M, Wei R, Andrews HF, Acosta EP, Bell KL, Pelton GH, Deliyannides D, Perrin AC, Caccappolo E, Gershon AA, Prasad KM, Kreisl WC, Mintz A, Huey ED. Valacyclovir Treatment of Early Symptomatic Alzheimer Disease: The VALAD Randomized Clinical Trial. JAMA. 2025 Dec 17:e2521738. doi: 10.1001/jama.2025.21738. Online ahead of print. PMID 41405855
- [Derived] Devanand DP, Andrews H, Kreisl WC, Razlighi Q, Gershon A, Stern Y, Mintz A, Wisniewski T, Acosta E, Pollina J, Katsikoumbas M, Bell KL, Pelton GH, Deliyannides D, Prasad KM, Huey ED. Antiviral therapy: Valacyclovir Treatment of Alzheimer's Disease (VALAD) Trial: protocol for a randomised, double-blind,placebo-controlled, treatment trial. BMJ Open. 2020 Feb 6;10(2):e032112. doi: 10.1136/bmjopen-2019-032112. PMID 32034019

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in 3 U.S. academic sites: Columbia University, New York University, and Banner Health.
Groups:
- Valacyclovir: 60 participants were assigned to receive valacyclovir for 78 weeks. Oral valacyclovir was distributed in 500 mg caplets. Participants took 8 caplets per day, 4 caplets in the morning and 4 caplets in the evening.
- Placebo: 60 participants were assigned to receive placebo for 78 weeks. The oral placebo (sugar pill) was matched in appearance to valacyclovir and distributed in 500 mg caplets. Participants took 8 caplets per day divided into 4 caplets in the morning and 4 caplets in the evening.
Period: Overall Study
Arm/Group | Valacyclovir | Placebo
Started | 60 | 60
Completed | 44 | 47
Not Completed | 16 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valacyclovir | Placebo | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (8.8) | 71.6 (8.6) | 71.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 31 | 66
  Male | 25 | 29 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 44 | 41 | 85
  Black non-Hispanic | 4 | 8 | 12
  Hispanic | 9 | 10 | 19
  Asian | 3 | 0 | 3
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120
ADAS-Cog11 [Mean (Standard Deviation); unit: units on a scale] — The Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog11) is an 11-item assessment used to assess the severity of cognitive dysfunction in Alzheimer's disease. The full range is 0 to 70, where a higher score indicates worse cognition. This is a neuropsychological test administered in person by a trained research staff member.
  units on a scale | 20.6 (6.6) | 19.2 (7.6) | 19.9 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer's Disease Assessment Scale - Cognition (ADAS-COG11, Modified Version) Score
Description: The modified ADAS-COG11 is a neuropsychological test used to measure the severity of cognitive dysfunction in Alzheimer's disease. The full range is 0 to 70, where a higher score indicates worse cognition.
Time Frame: Baseline, Week 78
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Valacyclovir | Placebo
Number analyzed (Participants) | 60 | 60
score on a scale
  Baseline | 20.6 (6.6) | 19.2 (7.6)
  78 weeks | 30.2 (13.9) | 25.3 (11.8)
Statistical Analysis 1: Comparison: Valacyclovir vs Placebo; Null hypothesis: there is no difference in change in ADAS-Cog11 between valacyclovir and placebo treatment. A sample size of 130 participants (65 per arm) was originally projected to detect Cohen's d of 0.50 with 80% power at 5% significance level. Recruitment target was reduced to 120 participants due to pandemic-related recruitment delays and required study completion within the extended funding timeline. For n=120, the minimum detectable effect size increased slightly to Cohen's d of 0.52; Test type: Superiority — Linear mixed-effects models (LMM) were used to assess the treatment effects on the outcome with change score from baseline as the dependent variable and treatment, study time point, and their interaction as predictors, adjusting for baseline value of the outcome; p < 0.05, Mixed Models Analysis — Not adjusted for multiple comparisons; Adjusting for baseline value of ADAS-Cog11; Mean Difference (Final Values) = 3.91, 95% CI 2-sided [1.03 to 6.80]

2. Secondary Outcome: Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) Score
Description: ADCS-ADL is a caregiver-reported scale to assess a patient's ability to perform everyday tasks. The full score range 0 to 78, with higher scores indicating better functioning.
Time Frame: Baseline, Week 78
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Valacyclovir | Placebo
Number analyzed (Participants) | 60 | 60
score on a scale
  Baseline | 65.8 (10.5) | 65.6 (11.4)
  Week 78 | 52.4 (20.9) | 54.3 (19.8)

3. Secondary Outcome: Total 18F-Florbetapir Brain Uptake
Description: 18F-Florbetapir PET imaging will show amyloid accumulation in a sum of six ROIs (Region of Interest) (cerebellar reference) that show increased uptake in AD: medial orbital frontal, anterior cingulate, parietal, temporal, posterior cingulate, precuneus. The full range is approximately 0 to 4 SUVR (Standardized Uptake Value Ratio), with higher SUVR indicating more amyloid.
Time Frame: Baseline, Week 78
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Valacyclovir | Placebo
Number analyzed (Participants) | 60 | 60
SUVR
  Baseline | 1.57 (0.37) | 1.57 (0.41)
  Week 78 | 1.63 (0.35) | 1.60 (0.41)

4. Secondary Outcome: Total 18F-MK-6240 Temporal Lobe Brain Uptake
Description: 18F-MK-6240 tau PET imaging will show tau accumulation, SUVR: average of medial temporal regions (amygdala, hippocampus, entorhinal, parahippocampus) with cerebellar reference. The full range is approximately 0 to 5 SUVR, with higher SUVR indicating more tau accumulation.
Time Frame: Baseline, Week 78
Population: MK-6240 PET imaging was funded by a grant supplement after the study began and therefore the number of participants for this component was less than the total sample.
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Valacyclovir | Placebo
Number analyzed (Participants) | 47 | 49
SUVR
  Baseline | 2.18 (0.82) | 1.91 (0.88)
  Week 78: number analyzed (Participants) | 24 | 31
  Week 78 | 2.32 (0.79) | 1.90 (0.89)

ADVERSE EVENTS:
Time Frame: 78 weeks
Description: Adverse events information was reported by the participant or informant without a specific scale being administered.
Arm/Group | Valacyclovir | Placebo
All-Cause Mortality (participants affected / at risk) | 2/60 | 2/60
Serious Adverse Events (participants affected / at risk) | 14/60 | 11/60
Other Adverse Events (participants affected / at risk) | 11/60 | 8/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valacyclovir (N=60) | Placebo (N=60)
Seizure, confusion (Nervous system disorders) | 2 (2) | 0 (0)
Respiratory distress, pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5)
Falls (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Kidney failure (Renal and urinary disorders) | 3 (3) | 1 (1)
Cardiac (Cardiac disorders) | 3 (3) | 3 (3)
nausea, abdominal pain, diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valacyclovir (N=60) | Placebo (N=60)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2) — 3 participants on valacyclovir and 2 participants on placebo developed nausea.
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Cardiovascular (Cardiac disorders) | 2 (2) | 2 (2)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations included the small sample size. The COVID-19 pandemic contributed to a dropout rate of 24%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-07-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT03282916/Prot_000.pdf
  • Statistical Analysis Plan (2025-07-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT03282916/SAP_001.pdf